CLINICAL TRIAL: NCT02747017
Title: An International Prospective Observational Study to Assess the Characteristics and Outcomes of Post-transplant Patients Treatment for C. Difficile Infections
Brief Title: Observational Study of C. Diff in Post-Transplant Patients
Acronym: CDIFF
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: International Network for Strategic Initiatives in Global HIV Trials (INSIGHT) (Network); Merck Sharp & Dohme LLC (Industry); Astellas Pharma Inc (Industry); Copenhagen HIV Programme (Other Government); Medical Research Council (Other Government); Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 1605M87565
Record Dates: First submitted 2016-04-12; First posted 2016-04-21 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Clostridium Difficile
Keywords: transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, stool
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CDI patients: Adults with a first episode of CDI within 2 years after solid-organ or stem-cell transplant.

SUMMARY:
The primary objective of this observational study is to estimate the 90-day response rates to treatment for a first episode of C. difficile infections (CDI) in adult transplant recipients.

DETAILED DESCRIPTION:
The primary objective of this observational study is to estimate the 90-day response rates to treatment for a first episode of C. difficile infections (CDI) in adult transplant recipients. This includes treatment success, recurrence, and complications in a prospectively followed cohort of solid organ and hematopoietic stem cell transplant patients. Patients who develop CDI within 2 years after transplantation will be enrolled and followed prospectively for 90 days after enrollment. Specimens of stool and serum collected within 48 hours of initiation of treatment will be stored locally for future epidemiologic studies to examine the immunologic and microbiologic risk factors for relapse and treatment failure, as well as complications of CDI in the transplant population. Response rates will be classified by organ type, hematopoietic stem cell transplant typ, treatment regimen, and immunosuppressive regimen.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Signed informed consent
* Transplant recipient (solid organ, stem cells, or bone marrow) within past 2 years
* Currently diagnosed with first CDI after transplant, defined by (1) presence of diarrhea (at least 3 loose stools within a 24-hour period), AND (2) detection of C. difficile cytotoxin in stools by cytotoxin assay, or toxigenic culture, or polymerase chain reaction (PCR) testing for toxin, or enzyme immunoassay, or endoscopic presence of pseudomembranes with the detection of C. difficile in tissue biopsies

Exclusion Criteria:

* Previous episode of CDI anytime after transplant
* Current treatment for another infectious cause of diarrhea (bacterial, viral, or parasitic) at the time of the current CDI diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with a first episode of CDI within 2 years post solid-organ or stem-cell transplant.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2016-08-22 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Response to antibiotic treatment for CDI: clinical cure | 90 days
  The planned first course of CDI treatment was completed with resolution of symptoms or less than 3 loose stools per day for at least two consecutive days maintained until end of treatment and two days after treatment course ended.
Response to antibiotic treatment for CDI: sustained clinical cure | 90 days
  Clinical cure achieved and maintained for 40 days post treatment initiation without recurrences, complications, ICU with CDI, or death as defined below
Response to antibiotic treatment for CDI: global cure | 90 days
  Clinical cure achieved and maintained for 90 days post treatment initiation without recurrences, complications, including ICU with CDI, or death as defined below.
Response to antibiotic treatment for CDI: relapse | 90 days
  A new episode of CDI after clinical cure and within 4 weeks after treatment initiation.
Response to antibiotic treatment for CDI: reinfection | 90 days
  A new episode of CDI after clinical cure and beyond 4 weeks after treatment initiation
Response to antibiotic treatment for CDI: complications | 90 days
  The study will collect the incidence of specific complications as assessed by the site investigator: perforation of the colon; development of toxic megacolon; need for abdominal surgery related to CDI; transfer to the ICU with CDI; death from CDI-related cause.

SECONDARY OUTCOMES:
Describe patients who are successfully treatment for CDI | 90 days
  Patients will be described by demographics (age, race, sex), type of transplant received, specific treatment for CDI, and the strain of C. difficile with which they were infected.
Describe differences in antibiotic regimens and other CDI treatments across geographic regions (US, Europe, South America) | 90 days
All-cause mortality | 90 days
Response to treatment for CDI (as defined above) by treatment regimen | 90 days
Response to treatment for CDI (as defined above) by type of transplant (solid organ vs. hematopoietic/stem cell) | 90 days
Assay differences across sites | 90 days
  Describe assays used to detect C. difficile organisms and toxin in stool by site at which participants are enrolled.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Molina, MD, Study Chair — Hôpital Saint-Louis, Service de Maladies Infectieuses
Locations (9):
- United States (4):
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina
- CHIP, Department of Infectious Diseases, Section 2100, Copenhagen, Denmark
- Klinik I fur Innere Medizin der Universitat zu Koln, Studienburo fur Infektiologie u. HIV, Cologne, Germany
- Spain (2):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Doce de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: INSIGHT network website, CDIFF home page — http://insight.ccbr.umn.edu/i07/
- Available data/document: Study Protocol — http://insight.ccbr.umn.edu/official_documents/CDIFF/protocol_documents/I7-Protocol.pdf